CLINICAL TRIAL: NCT06243887
Title: Implementing Enhanced Recovery After Surgery (ERAS) Protocol in Patients Undergoing Minimal Invasive Esophagectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Khaled Hassaan Mohamed Hussein, assistant lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: Minimal invasive esophegectomy
Record Dates: First submitted 2023-12-19; First posted 2024-02-06 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Esophageal Diseases; Esophagostomy Complication
MeSH Terms: conditions — Esophageal Diseases | interventions — Enhanced Recovery After Surgery; Clinical Protocols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional group (Other): patients of minimally invasive esophagectomy with standard of care approaches
  Interventions: Other: standard of care approaches in minimal invasive esophagectomy
- ERAS group (Other): patients of minimally invasive esophagectomy with enhanced recovery after surgery protocol
  Interventions: Other: Enhanced Recovery After Surgery (ERAS) protocol in minimal invasive esophagectomy

INTERVENTIONS:
Other: Enhanced Recovery After Surgery (ERAS) protocol in minimal invasive esophagectomy — Enhanced Recovery After Surgery (ERAS) refers to patient-centered, evidence-based, multidisciplinary team developed pathways for a surgical specialty and facility culture to reduce the patient's surgical stress response, optimize their physiologic function, and facilitate recovery.
  Arms: ERAS group
Other: standard of care approaches in minimal invasive esophagectomy — standard of care approaches other than ERAS
  Arms: Conventional group

SUMMARY:
Detect impact of enhanced recovery after surgery (ERAS) on the outcomes of oesophageal surgery .

DETAILED DESCRIPTION:
esophagectomy for both malignant and benign disease has been identified as a particularly complex surgical procedure due to documented high levels of peri-operative morbidity and mortality.

A comprehensive review of complications associated with the esophagectomies performed in high-volume esophageal units utilizing a standardized format for documenting complications and quality measures has confirmed an overall complication rate of 59 % with 17.2% of patients sustaining complications of IIIb or greater utilizing the Clavien-Dindo severity grading system. post-operative complications include high rate of anastomotic leakage , pulmonary infection ,thoracic duct injury , voice changes , breathlessness ,long hospital stay.

These outcomes accentuate the need for providing an enhanced recovery after surgery standardized format for esophagectomy which can be routinely applied and audited to improve international outcomes. though ERAS lacking randomized control trials

ELIGIBILITY:
Inclusion Criteria:

* 1) first detected and endoscopically confirmed esophageal cancer; 2)preoperative evaluation showed no distant metastases and suitable for MIE; 3preoperative clinical stage of I to III

Exclusion Criteria:

* 1) patients had a history of thoracic or abdominal surgery; 2)patients were IV to VI in the American Society of Anesthesiologists (ASA) physical status classification system; 3)patients had other malignancies; 4)patients had missing clinical data

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Enhanced recovery after surgery (ERAS) | average 2 years
  Detect impact of enhanced recovery after surgery on the outcomes of oesophageal surgery concerning
  1. time to out-of-bed activity
  2. time to first flatus
  3. time to liquid diet
  4. postoperative hospital stay
  5. ICU length of stay
  6. ICU length of stay
  7. in-hospital mortality
  8. incidence of various postoperative complications

SECONDARY OUTCOMES:
Enhanced recovery after surgery (ERAS) | average 2 years
  Detect impact of enhanced recovery after surgery on the outcomes of oesophageal surgery concerning
  1)postoperative chest drainage volume

REFERENCES:
- [Background] Puccetti F, Klevebro F, Kuppusamy M, Han S, Fagley RE, Low DE, Hubka M. Analysis of Compliance with Enhanced Recovery After Surgery (ERAS) Protocol for Esophagectomy. World J Surg. 2022 Dec;46(12):2839-2847. doi: 10.1007/s00268-022-06722-7. Epub 2022 Sep 22. PMID 36138318
- [Background] Shen Y, Chen X, Hou J, Chen Y, Fang Y, Xue Z, D'Journo XB, Cerfolio RJ, Fernando HC, Fiorelli A, Brunelli A, Cang J, Tan L, Wang H; Written on behalf of the AME Thoracic Surgery Collaborative Group. The effect of enhanced recovery after minimally invasive esophagectomy: a randomized controlled trial. Surg Endosc. 2022 Dec;36(12):9113-9122. doi: 10.1007/s00464-022-09385-6. Epub 2022 Jun 30. PMID 35773604